CLINICAL TRIAL: NCT03686358
Title: Evaluation of Renal Angioplasty on Atherosclerotic Stenosis Since 2010
Acronym: PARAS
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3069
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Renal Angioplasty on Atherosclerotic Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Renal artery angioplasty — Patients meeting the inclusion criteria were selected from the medical records of renal angioplasty performed at the Rennes University Hospital between 01/01/2010 and 12/31/2013. Each selected patient will receive a notice by mail of information. In the absence of opposition from them within a two weeks, the processing of their data will begin :
  * Evaluation of the results at 3 years of renal angioplasty on atherosclerotic stenosis performed at Rennes University Hospital
  * Evaluation of indications of renal angioplasty on stenosis atherosclerosis performed after 2009 at Rennes University Hospital
  * Identification of prognostic factors

SUMMARY:
The interest of renal angioplasty in the nosological framework of atherosclerotic stenosis has been significantly challenged by STAR and ASTRAL clinical trials in 2009, confirmed by the CORAL study in 2014.

These studies did not show any benefit of the gesture on renal function, morbidity and cardiovascular mortality or the tension control. The aim of the study is to evaluate renal angioplasty on atherosclerotic stenosis.

DETAILED DESCRIPTION:
Previous studies did not concern the indication of renal angioplasty in some high-risk situations, such as malignant or resistant renal vascular hypertension, OAP (Acute pulmonary oedema) flash or acute renal failure of ischemic origin.

There is no work in the literature that has studied retrospectively the evolution of angioplasty practices renal artery disease on atherosclerotic stenosis since 2009, nor their remote results of the gesture.

ELIGIBILITY:
Inclusion Criteria:

* OAP flash: hospitalization for Acute congestive heart failure without any other identified etiology than renal artery stenosis
* Resistant arterial hypertension under treatment including a diuretic
* Acute renal failure or ischemic renal failure quickly progressive
* Radiological criteria: renal ischemia visualized at arterial time of angio-CT or renal angio-MRI

Exclusion Criteria:

* Renal transplant patients
* Patients with another etiology of secondary hypertension, including fibro-muscular dysplasia of renal artery
* Restenosis on stent, angioplasty of accessory renal artery
* Patients subject to legal protection (safeguard of justice, guardianship) and persons deprived of liberty
* Patients objecting to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having undergone renal arterial angioplasty on atherosclerotic stenosis between 01/01/2010 and 12/31/2013 at Rennes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Composite endpoint at 3 years | The inclusion day
  Composite endpoint at 3 years :
  * Cardiovascular or renal mortality,
  * Initiation of a renal replacement therapy or estimated glomerular filtration rate decrease of more than 50%, Cardiovascular morbidity: hospitalization for congestive heart failure, myocardial infarction, myocardium, stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry FROUGET, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, Brittany Region, France